CLINICAL TRIAL: NCT00640783
Title: Effect of a Mediterranean-Style Diet on Endothelial Dysfunction and Markers of Vascular Inflammation in the Metabolic Syndrome
Brief Title: Mediterranean Diet and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Dario Giugliano, MD, PhD, Department of Geriatrics and Metabolic Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DGMM/06/2000
Record Dates: First submitted 2008-03-04; First posted 2008-03-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Mediterranean diet; Inflammatory markers; Endothelial function
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Mediterranean diet
  Interventions: Behavioral: Mediterranean diet
- 2 (Active Comparator): Control diet
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Mediterranean diet — The dietary advice was tailored to each patient on the basis of 3-day food records. The recommended composition of the dietary regimen was as follows: carbohydrates, 50% to 60%; proteins, 15% to 20%; total fat, less than 30%; saturated fat, less than 10%; and cholesterol consumption, less than 300 mg per day. Moreover, patients were advised to consume at least 250 to 300 g of fruits, 125 to 150 g of vegetables, and 25 to 50 g of walnuts per day; in addition, they were also encouraged to consume 400 g of whole grains (legumes, rice, maize, and wheat) daily and to increase their consumption of olive oil.
  Arms: 1
Behavioral: Control — Patients consuming the control diet were given general oral and written information about healthy food choices at baseline and at subsequent visits but were offered no specific individualized program. However, the general recommendation for macronutrient composition of the diet was similar to that for the intervention group (carbohydrates, 50%-60%; proteins, 15%-20%; and total fat, <30%).
  Arms: 2

SUMMARY:
The metabolic syndrome has been identified as a target for dietary therapies to reduce risk of cardiovascular disease; however, the role of diet in the etiology of the metabolic syndrome is poorly understood. To assess the effect of a Mediterranean-style diet on endothelial function and vascular inflammatory markers in patients with the metabolic syndrome

Randomized, single-blind trial conducted from June 2001 to January 2004 at a university hospital in Italy among 180 patients (99 men and 81 women) with the metabolic syndrome, as defined by the Adult Treatment Panel III.

Patients in the intervention group (n = 90) were instructed to follow a Mediterranean-style diet and received detailed advice about how to increase daily consumption of whole grains, fruits, vegetables, nuts, and olive oil; patients in the control group (n = 90) followed a prudent diet (carbohydrates, 50%-60%; proteins, 15%-20%; total fat, <30%).

After 2 years, patients following the Mediterranean-style diet consumed more foods rich in monounsaturated fat, polyunsaturated fat, and fiber and had a lower ratio of omega-6 to omega-3 fatty acids. Total fruit, vegetable, and nuts intake (274 g/d), whole grain intake (103 g/d), and olive oil consumption (8 g/d) were also significantly higher in the intervention group (P<.001). The level of physical activity increased in both groups by approximately 60%, without difference between groups. Mean body weight decreased more in patients in the intervention group (-4.0 kg) than in those in the control group (-1.2 kg) (P<.001). Compared with patients consuming the control diet, patients consuming the intervention diet had significantly reduced serum concentrations of hs-CRP (P = .01), IL-6 (P = .04), IL-7 (P = 0.4), and IL-18 (P = 0.3), as well as decreased insulin resistance (P<.001). Endothelial function score improved in the intervention group but remained stable in the control group. At 2 years of follow-up, 40 patients in the intervention group still had features of the metabolic syndrome, compared with 78 patients in the control group (P<.001).

A Mediterranean-style diet might be effective in reducing the prevalence of the metabolic syndrome and its associated cardiovascular risk.

DETAILED DESCRIPTION:
Patients consuming the intervention diet were given detailed advice about the usefulness of the experimental diet. Through a series of monthly small-group sessions, intervention patients received education in reducing dietary calories (if needed), personal goal-setting, and self-monitoring using food diaries. Behavioral and psychological counseling was also offered. The dietary advice was tailored to each patient on the basis of 3-day food records. The recommended composition of the dietary regimen was as follows: carbohydrates, 50% to 60%; proteins, 15% to 20%; total fat, less than 30%; saturated fat, less than 10%; and cholesterol consumption, less than 300 mg per day. Moreover, patients were advised to consume at least 250 to 300 g of fruits, 125 to 150 g of vegetables, and 25 to 50 g of walnuts per day; in addition, they were also encouraged to consume 400 g of whole grains (legumes, rice, maize, and wheat) daily and to increase their consumption of olive oil. Patients were in the program for 24 months and had monthly sessions with the nutritionist for the first year and bimonthly sessions for the second year. Compliance with the program was assessed by attendance at the meetings and completion of the diet diaries.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in the study, patients had to have 3 or more of the following criteria to meet the diagnosis of the metabolic syndrome, as defined by the Adult Treatment Panel III

Exclusion Criteria:

* Patients were excluded if they had cardiovascular disease, psychiatric problems, a history of alcohol abuse (alcohol consumption 500 g/wk in the last year), if they smoked, or if they took any medication.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2001-06; Primary Completion 2003-10 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function and vascular inflammatory markers | 2 years

SECONDARY OUTCOMES:
Resolution of metabolic syndrome | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD, PhD, Principal Investigator — Department of Geriatrics and Metabolic Diseases
Locations (1):
- Department of Geriatrics and Metabolic Diseases, Naples, Italy

REFERENCES:
- [Result] Esposito K, Marfella R, Ciotola M, Di Palo C, Giugliano F, Giugliano G, D'Armiento M, D'Andrea F, Giugliano D. Effect of a mediterranean-style diet on endothelial dysfunction and markers of vascular inflammation in the metabolic syndrome: a randomized trial. JAMA. 2004 Sep 22;292(12):1440-6. doi: 10.1001/jama.292.12.1440. PMID 15383514